CLINICAL TRIAL: NCT01653873
Title: to Compare the Efficacy of Parameters From Different Imaging Modality in Predicting the Risk of Future Vertebral Compression Fracture in Osteoporotic Patients.
Brief Title: Imaging Parameters to Predict Future Vertebral Fracture in Osteoporosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Chairman, National Taiwan University Hospital
Other Study IDs: 201202077RIC
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Osteoporosis; Fracture
Keywords: fracture; vertebral column; osteoporosis; predictor; vertebroplasty
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
After vertebroplasty, many patients will suffer from 2nd fracture in the vertebral column. With analyzing of the images done right after the 1st vertebroplasty, we can define the parameters from different imaging and they can be predictors of the future fracture.

DETAILED DESCRIPTION:
Vertebroplasty is considered one of the alternatives for the treating of spine compression fracture associated with pain especially for those patients with osteoporosis. However, after vertebroplasty, the compliance of the bone becomes stronger than the adjacent vertebrae that is not treated. So there is always a consideration of future fracture of the adjacent vertebral bodies after vertebroplasty done on certain body. In this study, we try to follow the patients (5 years) to see if the adjacent vertebral bodies are prone to have fracture than the others away from the site of vertebroplasty.Then we try to find out the image biomarkers to predict the future fracture in the vertebral bodies. The should be done with CT scan raw data, analysis with different algorithms.

Inclusion criteria; patients with osteoporosis and receiving vertebroplasty and with secondary fracture occurring in other spine exclusion criteria: No second vertebral body fracture occurred. Primary measurement: the time and location of the 2nd fracture secondary measurement: the imaging biomarkers from CT scan.

ELIGIBILITY:
Inclusion Criteria:

* All the patients received vertebroplasty treatment between 2005.01-2011.12 with 2nd fracture in the vertebral column.

Exclusion Criteria:

* No image available

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all the patients received vertebroplasty treatment between 2005.01-2011.12
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
fracture | 5 years
  2nd fracture within 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hon-Man Liu, MD, MBA, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Ito M, Ikeda K, Nishiguchi M, Shindo H, Uetani M, Hosoi T, Orimo H. Multi-detector row CT imaging of vertebral microstructure for evaluation of fracture risk. J Bone Miner Res. 2005 Oct;20(10):1828-36. doi: 10.1359/JBMR.050610. Epub 2005 Jun 20. PMID 16160740